CLINICAL TRIAL: NCT03879395
Title: Surgery for Gastrointestinal Metastases of Malignant Melanoma - a Single Center Retrospective Cohort Study
Acronym: SurgMelMet
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate Professor, Senior Consultant Surgeon, Sahlgrenska University Hospital
Other Study IDs: SurgMelMet
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Melanoma Stage Iv; Melanoma Metastatic; Abdominal Tumor
Keywords: melanoma; abdominal metastasis; metastasectomy; tumor resection; M1c
MeSH Terms: conditions — Melanoma; Abdominal Neoplasms | interventions — Metastasectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients with stage IV malignant melanoma with abdominal metastasis (M1c) that underwent abdominal surgery with metastasectomy during the study period.
  Interventions: Procedure: Abdominal surgery with metastasectomy

INTERVENTIONS:
Procedure: Abdominal surgery with metastasectomy — Emergency or elective surgery on indications related to abdominally metastasized malignant melanoma

SUMMARY:
The aim is to conduct a single centre retrospective study of all patients with stage IV melanoma that underwent surgery for metastases at Sahlgrenska University Hospital between 2010-01-01 and 2018-12-31. Pre- and postoperative data will be collected from digital medical records, the Swedish Cancer Registry, the Swedish Cause of Death Register as well as from the national Swedish cancer patient database (INCA). If needed, patient records will be collected from other hospitals. Results will be presented in written format as a summary and analysis of the characteristics of the cases operated on during the inclusion period.

The aim is to identify predictive and prognostic factors for outcome and complications in the surgical treatment of stage IV metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy verified stage IV malignant melanoma, stage M1c.
* Having undergone surgery with metastasectomy of melanoma tumors.

Exclusion Criteria:

* retroperitoneal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominally metastasized malignant melanoma stage IV.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | December 2018
  Overall survival

SECONDARY OUTCOMES:
Complications according to Clavien-Dindo within 90 days. | 90 days
  Complications according to Clavien-Dindo within 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data to be made available upon request.

REFERENCES:
- [Derived] Holmberg CJ, Alwan G, Ny L, Olofsson Bagge R, Katsarelias D. Surgery for gastrointestinal metastases of malignant melanoma - a retrospective exploratory study. World J Surg Oncol. 2019 Jul 12;17(1):123. doi: 10.1186/s12957-019-1663-z. PMID 31299988